CLINICAL TRIAL: NCT04834388
Title: Anakinra in Cerebral Haemorrhage to Target Secondary Injury Resulting From Neuroinflammation - a Phase II Clinical Trial
Brief Title: Studying Anakinra to Reduce Secondary Brain Damage After Spontaneous Haemorrhagic Stroke
Acronym: ACTION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL76607.091.21
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: PROBE design
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anakinra High dose (Experimental): 500mg i.v. loading dose, followed by continuous iv infusion with 2mg/kg/h over 3 days
  Interventions: Drug: Anakinra
- Anakinra Low dose (Experimental): 100mg s.c. loading dose, followed by subcutaneous administration of 100mg twice daily for 3 days.
  Interventions: Drug: Anakinra
- Standard care (No Intervention): Standard care group

INTERVENTIONS:
Drug: Anakinra — Anakinra treatment is started within 8 hours of symptom onset
  Other Names: Kineret
  Arms: Anakinra High dose; Anakinra Low dose

SUMMARY:
The goal of this clinical trial] is to determine if anakinra can ameliorate the formation of perihaematomal oedema in patients with spontaneous intracerebral haemorrhage (ICH). The main aims are:

* To determine the effect of high-dose versus low-dose anakinra compared to standard medical management on perihaematomal oedema formation in the first week after ICH.
* Determine the safety profile of anakinra in these patients
* Study the effect of anakinra treatment on inflammation markers, blood-brain-barrier permeability and functional outcome.

Researchers will compare treatment with anakinra for three days, in either a low or high dose, with standard medical care after ICH. Participants will:

* Be randomized to receive anakinra during three days, or receive standard medical care
* Undergo a MRI scan seven days after their ICH
* Take part in a telephone interview their functional performance three months later.

DETAILED DESCRIPTION:
Spontaneous intracerebral haemorrhage (sICH) is the deadliest stroke subtype yearly affecting over 6000 patients in the Netherlands. Treatment options are very limited. Inflammation plays a vital role in the development of sICH-related secondary brain injury (SBI). Within 4 hours after sICH onset, blood components and thrombin induce the release of cytokines and other inflammatory molecules, with subsequent microglial activation, blood brain barrier (BBB) damage and the formation of perihaematomal oedema (PHO). Among the released cytokines, interleukin 1 beta (IL-1β) has a pivotal role. Recombinant human interleukin-1 receptor antagonist (IL-1Ra, anakinra) effectively antagonizes IL-1β through competitive binding to the IL-1 receptor. Anakinra is available for treatment of rheumatoid arthritis, other inflammatory diseases and has been studied in acute sepsis. We hypothesize that anakinra safely reduces SBI after sICH, and that its effect is dose-dependent.

Objective: To determine the effect of high-dose versus low-dose anakinra compared to standard medical management on oedema extension distance (OED) determined with MRI on day 7±1. Second, to study the safety profile of anakinra. Furthermore, to assess its effect on 1) serum inflammatory markers IL-1β, IL-6, hsCRP, neutrophil and total white blood cell counts at day 1, 3 and 7 compared to baseline; 2) dynamic contrast enhanced (DCE-) MRI measurement of BBB transfer constant (Ktrans) on day 7±1, and; 3) to estimate an effect on functional outcome in patients with sICH.

Study design: Multicentre, prospective, randomized, three-armed (1:1:1) trial with open label treatment and blinded end-point assessment (PROBE design) .

Study population: 75 patients with supratentorial sICH admitted within 8 hours after symptom onset.

Intervention: Patients will receive anakinra in either a high dose (loading dose 500mg i.v., followed by infusion with 2mg/kg/h over 3 days; n=25) or in a low dose (loading dose 100mg s.c.., followed by subcutaneous administration of 100mg twice a day for 3 days; n=25), started within 8 hours of symptom onset. The control group (n=25) will receive standard medical management.

Main study parameters/endpoints: Primary objective is to test whether anakinra reduces subacute perihaematomal oedema after sICH, measured as OED on MRI at day 7±1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Supratentorial non-traumatic ICH confirmed by CT, without a confirmed causative lesion on admission CT-angiography (e.g. aneurysm, AVM, DAVF, cerebral venous sinus thrombosis) or other known underlying lesion (e.g. tumour, cavernoma);
3. Minimal intracerebral haemorrhage volume of 10 mL;
4. Intervention can be started within 8 hours from symptoms onset;
5. Patient's or legal representative's informed consent.

Exclusion Criteria:

1. Severe ICH, unlikely to survive the first 72 hours (defined as Glasgow Coma Scale score < 6 at time of consent);
2. Confirmed or suspected haemorrhagic transformation of an arterial or venous infarct;
3. Planned neurosurgical haematoma evacuation;
4. Severe infection at admission, requiring antibiotic treatment;
5. Known active tuberculosis or active hepatitis;
6. Use of immunosuppressive or immune-modulating therapy at admission (see 15.1 Appendix A);
7. Neutropenia (Absolute Neutrophil Count (ANC) <1.5 x 109/L );
8. Pre-stroke modified Rankin Scale score ≥ 3;
9. Pregnancy or breast-feeding;
10. Standard contraindications to MRI (see 15.2 Appendix B);
11. Known prior allergic reaction to gadolinium contrast or one of the constituents of its solution for administration;
12. Known allergy to anakinra or other products that are produced by DNA technology using the micro-organism E. coli;
13. Live vaccinations within the last 10 days prior to this ICH;
14. Severe renal impairment (eGFR <30ml/min/1.73m)
15. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perihematomal oedema | 7 days after ICH onset
  Measured as Oedema Extension Distance (OED/EED)

SECONDARY OUTCOMES:
Adverse events of special interest (AESI) and serious adverse events (SAE) | 90 days
  Number of events in the control group versus the treatment groups
Blood brain barriere leakage | 7 days
  Measured as Ktrans on DCE-MRI
Levels of serum inflammatory markers (IL-1β, IL-6, hsCRP) | 7 days
  IL-1β, IL-6, hsCRP
Functional outcome | 90 days
  Ordinal shift in functional outcome on the modified rankin scale (mRS) (comparing the intervention group to the controls), assessed with the modified Rankin Scale (mRS) at 3 months. This is a six point scale in which a score of 0 means no symptoms at all, a higher score means more impairment, and a score of 6 means the participant is dead.

CONTACTS AND LOCATIONS:
Overall Officials: F.H.B.M. Schreuder, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cliteur MP, van der Kolk AG, Hannink G, Hofmeijer J, Jolink W, Klijn C, Schreuder F. Anakinra in cerebral haemorrhage to target secondary injury resulting from neuroinflammation (ACTION): Study protocol of a phase II randomised clinical trial. Eur Stroke J. 2024 Mar;9(1):265-273. doi: 10.1177/23969873231200686. Epub 2023 Sep 15. PMID 37713268
- See also: trial website — https://www.action-study.nl/